CLINICAL TRIAL: NCT05570396
Title: Long-term Follow-up on Childhood Adiposity After Randomized Controlled Lifestyle Interventions in Pregnancy - The FitKids Study
Brief Title: Long-term Follow-up on Childhood Adiposity - The FitKids Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Grete Katrine Teilmann, Clinical Associate Professor, Nordsjaellands Hospital
Other Study IDs: H-22018855
Record Dates: First submitted 2022-09-26; First posted 2022-10-06 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Child Obesity; Metabolic Syndrome; Physical Activity; Pregnancy Related; Child Health
MeSH Terms: conditions — Pediatric Obesity; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The FitKids study is a mother-child observational cohort study on obesity and metabolism in children three years of age. The study will follow up on the FitMum and FitBaby studies, conducted from 2018-2022. The children in FitKids are born by mothers who completed the FitMum study, a single-site three-armed RCT, targeting physical activity during pregnancy. 220 pregnant women were randomly assigned to one of three arms during pregnancy: structured supervised exercise training, motivational counselling supported by health technology, or a control group receiving standard treatment. From inclusion and until one-year post-partum, the women wore an activity tracker 24/7 providing important information about adherence to the prescribed intervention. The primary objective of the FitKids study is to investigate the effect of lifestyle interventions during pregnancy on body composition (fat percentage measured by dual energy x-ray absorptiometry) and risk of childhood obesity in off-springs.

The secondary objectives are to investigate the effect of lifestyle interventions during pregnancy on obesity-associated dys-metabolic traits and mental health in off-springs as well as to gain insight into presumed causal factors for overweight and obesity in children.

The investigators hypothesize that children of mothers, who during their participation in FitMum, received an intervention will have a healthier body composition expressed as a fat percentage within the normal range for a 3-year-old child compared to children of mothers in the control group.

DETAILED DESCRIPTION:
Worldwide obesity has nearly tripled since 1975. In 2020, 39 million children under the age of five were overweight or obese. In Denmark approximately 13% of children are overweight or severely overweight by the time they start school.

Overweight is generally defined as abnormal fat accumulation and obesity as excessive fat accumulation that may impair health. For children under five years of age, overweight is defined as weight-for-height greater than two standard deviations above World Health Organization (WHO) Child Growth Standards median. Obesity is defined as weight-for-height greater than three standard deviations above the WHO Child Growth Standards median. Childhood obesity is associated with an increased risk of adult obesity, type 2 diabetes, metabolic syndrome, early death and reduced mental health. The large scale of obesity and the serious health problems associated with it calls for more knowledge within the field to prevent children from becoming overweight.

Body growth, physical activity, diet, and mental health are focus areas with respect to prevention and treatment of childhood obesity. Current knowledge about both pre- and postnatal factors indicates that being exposed to an adverse fetal environment, including maternal obesity, enhances propagation of obesity and associated cardiometabolic comorbidities, including type 2 diabetes. Still, the evidence is inconsistent and leaves most questions unanswered.

Many studies have found strong associations between maternal BMI and their child's BMI. One study showed distinct differences between associations of child BMI with maternal BMI compared to paternal BMI at birth but with the difference between associations diminishing over time. Another study showed associations between maternal pre-pregnancy BMI and child BMI at age five - six years of age. Given this it seems reasonable to suggest that the intrauterine environment is likely associated with the growth trajectory of the young child.

It is known that intrauterine exposure to diabetes and size at birth are risk factors for developing type 2 diabetes mellitus later in life, but several studies have also shown that children of mothers with obesity and overweight/obese children are at risk of having early markers of metabolic syndrome, i.e., increased insulin resistance, disturbed lipid profiles and high blood pressure.

Lifestyle interventions (physical activity and/or diet) in pregnant women have shown potential to reduce gestational weight gain and are associated with epigenetic changes in the child, potentially influencing the child's lean mass and early growth. However, in a recent metanalysis, prenatal lifestyle interventions were not shown to influence childhood weight or growth, but adherence to prescribed interventions was not systematically considered in the included studies, and only few studies reported data on body composition and metabolism in the child. Therefore, previous studies may not capture more specific effects of prenatal exposures on child fat accretion. Detailed knowledge about maternal lifestyle during pregnancy, combined with advanced measurement of body-composition in children, may contribute to a deeper understanding of how peri- and postnatal factors influence risk of childhood obesity.

Body Mass Index (BMI) is strongly correlated with adiposity and the use of age and gender adjusted Body Mass Index (z-BMI) is a crude approximation of excess fat mass. However, BMI z-scores may in some children lead to misclassification of overweight or obesity. BMI has high specificity but low sensitivity to detect excess adiposity and fails to identify more than 25% of children with excess body fat percentage. To overcome the pitfalls associated with BMI, body composition can be measured. Body weight is the sum of fat-mass (FM) and fat-free mass (FFM), and body composition describes the relative proportion of fat-mass and fat-free mass in the body. Experts have not yet identified or agreed upon a definition of obesity that uses an absolute cut-off or threshold for increased body fat mass during childhood. Measuring fat percentage in children is challenging and requires the child to cooperate to the examinations. While Dual-energy X-ray Absorptiometry (DXA) scan is the gold standard, it is well recognized that compliance and cooperation in general is varying in younger children. Therefore, the use of other methods, e.g., air displacement plethysmography (BodPod), may be included in research of childhood obesity.

The FitKids-Cohort:

The FitKids study is a mother-child observational cohort study on health in children three years of age. The study will follow up on the FitMum (19) and FitBaby studies, conducted from 2018-2022.

The children in FitKids are born by mothers who completed the FitMum study, a single-site three-armed randomized controlled trial (RCT), targeting physical activity during pregnancy. 220 previously sedentary, healthy, pregnant women were included in the trial before gestational age (GA) week 15+0. The women had a BMI between 18.5-45 kg/m2 or a weight below 150 kg calculated from pre-pregnancy weight or first measured weight in pregnancy and all had a singleton pregnancy. Included women were randomly assigned to one of three arms during pregnancy: structured supervised exercise training (EXE), motivational counselling supported by health technology (MOT), or a control group receiving standard treatment (CON). From inclusion and until one-year post-partum, the women wore an activity tracker 24/7. This, providing important information about adherence to the prescribed intervention during pregnancy and their general level of activity both during pregnancy and one-year post-partum.

All children were invited to participate in The FitBaby study, which includes children who were born by FitMum participants and aims to evaluate the effects of maternal physical activity during pregnancy on health of the child at 12 months.

In FitMum and FitBaby, the effects of structured supervised exercise training and motivational counselling during pregnancy on physical activity level and health of mother and child are studied. 44% of FitMum participants were overweight or obese before conception and data regarding gestational weight gain as well as maternal weight during the first-year post-partum have been rigorously collected. The cohort is currently followed up during first year of life in the FitBaby study, and further follow-up in FitKids will add important knowledge about long term effects of the intra- and extrauterine environment on the risk of developing childhood overweight as well as growth, body composition, metabolism, and mental health.

The FitKids study is part of The LiP-TOP-Fit consortium consisting of three follow-up studies; LiPO Teen, a follow-up on the 14-15 year-old teenage offspring from the mothers of The Lifestyle in Pregnancy (LiP) study, TOP12, a follow-up on the 12 year old offspring from The Treatment of Obese Pregnant women (TOP) study and FitKids. Together with the FitKids follow up study the synergistic effect of the three follow-up programs in the LiP-TOP-Fit study entails a unique opportunity to understand long-term causal mechanisms of childhood obesity with possible substantially impact for future preventive strategies.

Expected outcomes:

The FitKids study provides a comprehensive assessment of childhood health, including whole body composition assessed by children anthropometric measures, dual energy x-ray absorptiometry (DXA) and BodPod as well as early markers of metabolic disease assessed by seven-day free-living continuous glucose monitoring, physical activity, blood samples and hair cortisol levels.

The children are uniquely well characterized using data from the biological mother during pregnancy and the child from birth until three years of age. Thus, allowing for assessment of fetal and postnatal programming effects. Hence, based on information from the FitMum and FitBaby studies the investigators can investigate early risk factors of later obesity. The longitudinal design allows for investigating trajectories and timing of risk factors, including level of physical activity, body composition and markers of metabolic disease e.g., insulin resistance. The investigators expect that the FitKids study will provide new insights in how body weight and composition in childhood track back to the intrauterine or early postnatal environment.

Expected significance of the project to deliver evidence of causal factors:

Building upon the RCT design in the FitMum study and the ongoing FitBaby study, the investigators seek to investigate causal relations between the pre- and postnatal environment and childhood health.

This can lead to the development of targeted interventions in the prevention of childhood obesity to be implemented at obstetric and/or paediatric departments

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from custody holders before any study related procedures are performed
2. The participants must be born by mothers participating in FitMum and born during the intervention period.

Exclusion Criteria:

There are no established exclusion criteria. If a potential participant suffers from a physical or mental illness the decision about participation will be decided together with the parent(s)/custody holder(s).

Ages: 36 Months to 47 Months | Sex: All
Age Groups: Child
Study Population: The research team is still in contact with the participants in FitMum and all children of mothers who completed FitMum will be invited to participate in the FitKids study. The FitMum cohort is 'loyal' as 81% of participants have remained in the study at least until delivery. Therefore, 178 children will be eligible for inclusion and receive an invitation to participate in the FitKids study. A subgroup of the children (n = 147) participated in or are currently participating in the FitBaby study at one year of age.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
fat percentage | Collection from October 2022 until June 2024
  fat percentage in three-year-old children of mothers who gave birth while still participating in the FitMum study measured by dual energy x-ray absorptiometry and Air Displacement Plethysmography technology

SECONDARY OUTCOMES:
BMI | Collection from October 2022 until June 2024
  Stature will be measured to the nearest 0.1 cm using a wall stadiometer, and body mass will be measured to the nearest 0.1 kg using a standard balance beam scale.
Waist-hip ratio | Collection from October 2022 until June 2024
  Waist, hip and abdominal circumference will be measured to the nearest 0.1 cm using a measuring tape.
Skinfolds | Collection from October 2022 until June 2024
  Triceps and subscapular skinfolds will be measured to the nearest millimeter with a skinfold caliper.
Blood pressure | Collection from October 2022 until June 2024
  Both systolic and diastolic blood pressure, will be measured after standard procedures. Before measuring the blood pressure, the child is to sit still on a chair with both feet flat on the ground or lie down for at least five minutes. The right cuff size is picked out by measuring the circumference of the upper arm midway between olecranon (elbow) and acromion (shoulder).
Heart rate | Collection from October 2022 until June 2024
  Heart rate will be measured when measuring the blood pressure after standard procedures. Before measuring the heart rate, the child is to sit still on a chair with both feet flat on the ground or lie down for at least five minutes.
Metabolic markers | Collection from October 2022 until June 2024.
  Plasma metabolites and hormones (e.g. glucose, total cholesterol, triglycerides, lipoproteins and Thyroid stimulating hormone) will be measured in blood samples collected by venipuncture after an overnight fast.
Epigenetics | Collection from October 2022 until June 2024.
  Epigenetic analyses will be perfomed on blood samples collected by venipuncture after an overnight fast.
Mesoscale analyses | Collection from October 2022 until June 2024.
  Mesoscale analyses will be performed on plasma from blood samples collected by venipuncture after an overnight fast.to detect protein and peptide concentrations.
Hair samples for cortisol levels | Collection from October 2022 until June 2024
  One hair sample from the child for measurements of cortisol levels.
Continuous glucose monitoring (CGM) | Collection from October 2022 until June 2024
  Fasting glucose, post prandial glucose values, glucose variability (7 days). Glucose metabolism will be measured through seven-day CGM (Dexcom G6). The CGM will provide information on fasting, prandial and postprandial glucose excursions as well as overall glycaemic variability
Physical activity behaviour | Collection from October 2022 until June 2024
  Physical Activity level will be measured in all participants by 7 days of 24-h activity tracking (Actigraphs GT3X+) placed around the wrist.
Sleep pattern | Collection from October 2022 until June 2024
  Sleep pattern will be measured in all participants by 7 days of 24-h activity tracking (Actigraphs GT3X+) placed around the wrist.
Food Frequency Questionnaire (FFQ) | Collection from October 2022 until June 2024
  Dietary habits will be assessed by the Food Frequency Questionnaire (FFQ) answered by a parent.
Ages & Stages Questionnaire (ASQ) | Collection from October 2022 until June 2024
  The psycho-motor development will be assessed by the Ages & Stages Questionnaire (ASQ) answered by a parent.
Strength and Difficulties Questionnaire (SDQ) | Collection from October 2022 until June 2024
  Mental health will be assessed by the Strength and Difficulties Questionnaire (SDQ) answered by a parent.
Pregnancy Physical Activity Questionnaire (PPAQ) | Collection from October 2022 until June 2024
  Physical activity in the birth mother will be assessed by the Pregnancy Physical Activity Questionnaire (PPAQ) answered by the birth mother.
Glucose challenge test | Collection from October 2022 until June 2024
  During CGM-recording, a standardized home setting non-invasive oral glucose challenge will be performed. The test runs over a period of two hours and the child must be fasting both before the test and not eat or drink during the test. The child will be offered 1 dl of sugar water containing 1.75 g glucose/kg; max 75g. Flavour in the form of sugar free soft drinks can be added to improve the taste. The sugar water is to be consumed in five min. Over the next two hours the caregiver must note the sensor glucose at time 0 minutes; 30 minutes and 120 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Grete K Teilmann, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Nordsjaellands Hospital, Hillerød, Denmark